CLINICAL TRIAL: NCT02249767
Title: Bioequivalence Study of Tretinoin Gel 0.05% to Brand Tretinoin Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spear Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tret.2014.10.01.14
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Generic Tretinoin (Active Comparator): Treatment of acne once daily over 12 weeks
  Interventions: Drug: Tretinoin
- Brand Tretinoin (Active Comparator): Treatment of Acne once daily over 12 weeks
  Interventions: Drug: Tretinoin
- Placebo Vehicle (Placebo Comparator): Treatment of acne once daily over 12 weeks
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: Tretinoin — Treatment of acne once daily in evening
  Other Names: Placebo

SUMMARY:
This was a double-blind, randomized, three-treatment, parallel study. Normal, healthy male and female children and adults (i.e., ages 12 to 40 years) with at least Grade 2 (i.e., mild severity) acne vulgaris were treated on the full face once daily for 84 days with the Tretinoin Gel 0.05%, Brand (tretinoin) Gel 0.05%, or Gel Vehicle. Acne lesions were graded by a single blinded observer at screening and at Weeks 0 (i.e., baseline), 2, 4, 8, and 12 at each location.

DETAILED DESCRIPTION:
This was a double-blind, randomized, three-treatment, parallel study conducted at three locations with a single investigator. Normal, healthy male and female children and adults (i.e., ages 12 to 40 years) with at least Grade 2 (i.e., mild severity) acne vulgaris were treated on the full face once daily for 84 days with the Tretinoin Gel 0.05%, Brand (tretinoin) Gel 0.05%, or Gel Vehicle. Acne lesions were graded by a single blinded observer at screening and at Weeks 0 (i.e., baseline), 2, 4, 8, and 12 at each location.

The assigned study treatment was self-applied topically once daily for 84 consecutive days. Scheduled study visits included:

* Visit 1 (Baseline Visit, Day 0)
* Visit 2 (First Interim Visit, Day 14)
* Visit 3 (Second Interim Visit, Day 28)
* Visit 4 (Third Interim Visit, Day 56)
* Visit 5 (Forth Interim Visit, Day 84)

A window of ± 4 days was considered acceptable for each scheduled visit following the Baseline Visit. Subjects were admitted into the study if they had a clinical diagnosis of acne vulgaris and if they met the inclusion/exclusion criteria. During the study visits, the following procedures were performed:

* Counts of inflammatory, non-inflammatory, and nodulocystic lesions
* The Investigator's Global Assessment (IGA)
* Assessment of application site reactions Safety was assessed by the monitoring of AEs and documenting signs and/or symptoms of application site reactions.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy male and female children and adults aged 12 to 40 years
* Written and verbal informed consent had to be obtained. Subjects aged 12 to 17 years, had to sign an assent for the study and a parent or a legal guardian had to sign the informed consent
* Women of childbearing potential had to be non-pregnant and non-nursing, and had to be willing to avoid pregnancy during the course of the study and during the menstrual cycle following completion of their participation in the study. Adequate contraception was defined as systemic birth control, such as oral contraceptives, for three months prior and implantable/injectable contraceptives (e.g., Norplant, intrauterine device [IUD]) for six months prior to study drug administration; or barrier methods, such as diaphragm plus spermicide or condom plus spermicide, consistently for at least 14 days prior to study drug administration; or abstinence.
* On the face, having ≥ 20 inflammatory (i.e., papules and pustules) and ≥ 25 non-inflammatory (i.e., open and closed comedones) lesions with ≤ 2 nodulocystic lesions (i.e, nodules and cysts), as per FDA Draft Guidance on Tretinoin, dated March 20
* Able to refrain from the use of all other topical acne medications or antibiotics during the treatment period
* Considered reliable and capable of understanding their responsibility and role in the study

Exclusion Criteria:

* Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis). Note: Eczema and psoriasis on the body are not exclusions.
* Subjects with active cystic acne as evidenced by more than 2 facial nodules. Nodules are defined as in 7.3.3 as: deep-seated in the skin (i.e., centered in the dermis or subcutis) and greater than 5 mm in diameter.
* More than 40 papules and/or pustules (inflammatory lesions).
* More than 60 open and/or closed comedones/milia (non-inflammatory lesions).
* Overall severity grade of less than 2 or greater than 4.
* History of allergy or hypersensitivity to tretinoin, retinoids, or any of the study medication ingredients.
* Significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hepatic, neurological, pancreatic, or renal disease.
* Use within 6 months prior to baseline of systemic retinoid (isotretinoin) treatment or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
* Oral contraceptives started or changed within 3 months prior to study initiation or planned to change during the study.
* Use on the face within 1 month prior to baseline of 1) cryodestruction or chemodestruction, 2) dermabrasion, 3) photodynamic therapy, 4) acne surgery, 5) intralesional steroids, or 6) x-ray therapy.
* Use within 1 month prior to baseline of 1) spironolactone, 2) systemic steroids, 3) systemic antibiotics, 4) systemic treatment for acne vulgaris (other than oral retinoids, which require a 6-month washout), or 5) systemic anti-inflammatory agents.
* Use within 2 weeks prior to baseline of 1) topical steroids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparations, 4) topical anti-inflammatory agents, or 5) topical antibiotics.
* Pregnant or breast-feeding.
* Serious psychological illness.
* Significant history (within the past year) of alcohol or drug abuse.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 574 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Barker, MD, Principal Investigator — Moore Clinical Research

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Generic Tretinoin | Brand Tretinoin | Placebo Vehicle
Started | 230 | 229 | 115
Completed | 222 | 220 | 107
Not Completed | 8 | 9 | 8
Not completed — Did not use medication | 8 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Tretinoin | Brand Tretinoin | Placebo Vehicle | Total
Number analyzed (Participants) | 222 | 220 | 107 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (7.06) | 20.1 (7.60) | 19.6 (7.31) | 20.0 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 131 | 64 | 319
  Male | 98 | 89 | 43 | 230
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 3 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 57 | 46 | 24 | 127
  White | 111 | 109 | 61 | 281
  More than one race | 50 | 60 | 16 | 126
  Unknown or Not Reported | 0 | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 222 | 220 | 107 | 549

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Baseline Acne Lesions at Week 12
Description: Percent change in baseline in inflammatory and non-inflammatory lesions at week 12.
Time Frame: Baseline and 12 weeks
Population: This is Per protocol population (PP) Analysis. Generic Tretinoin Intent to Treat (ITT) started 222- 22 excluded as not following protocol= 200 PP. Brand Tretinoin 220 ITT - 11 excluded not following Protocol=209 PP. Placebo 107 ITT - 7 excluded = 100 PP Percent change from baseline in acne lesions
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Generic Tretinoin | Brand Tretinoin | Placebo Vehicle
Number analyzed (Participants) | 200 | 209 | 100
Percent reduction | -32.34 (30.35) | -37.32 (28.81) | -26.38 (32.33)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Treatment related irritation
Arm/Group | Generic Tretinoin | Brand Tretinoin | Placebo Vehicle
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/229 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/230 | 0/229 | 0/115
Other Adverse Events (participants affected / at risk) | 49/230 | 46/229 | 26/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Tretinoin (N=230) | Brand Tretinoin (N=229) | Placebo Vehicle (N=115)
Irritation from Drug (Skin and subcutaneous tissue disorders) | 49 | 46 | 26 — Irritation from drug as expected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
With OK from Sponsor